CLINICAL TRIAL: NCT03943732
Title: Randomized Trial Measuring the Clinical Impact of the FilmArray® Pneumonia, a Prospective Interventional Trial
Brief Title: Trial Measuring the Clinical Impact of the FilmArray® Pneumonia Panel in Critically Ill
Acronym: FA-PNEU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: FA-PNEU; 2019/14MAR/124 (Other: CEHF)
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Pneumonia
Keywords: Pneumonia; Molecular Testing; Clinical impact; FilmArray Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: Open Randomized study, consecutive 2 weeks-period for observation group and study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Respiratory samples are treated according to routine laboratory testing : culture, immuno assays
- Intervention (Experimental): Respiratory samples are treated according to routine laboratory testing : culture, immuno assays AND molecular testing (FilmArray PNEU) of the endotracheal aspirate sample 24 hours a day.
  Interventions: Diagnostic Test: FilmArray Pneumonia

INTERVENTIONS:
Diagnostic Test: FilmArray Pneumonia — FilmArray Pneumonia testing of tracheal sample
  Arms: Intervention

SUMMARY:
The objective of this study is to measure how the use of Film-Array Pneumonia (FA-PNEU) on respiratory samples of adult patients suspected of acute care pneumonia in the intensive care unit of Saint-Luc University Hospital can accelerate / improve the initiation of the optimal antibiotic treatment.

DETAILED DESCRIPTION:
The main objective of this trial is to confirm/attest/prove the following statement:

The use of the FilmArray Pneumonia panel on respiratory samples of critically ill suspected with pneumonia, enables a faster microbiological pneumonia diagnosis and an improved therapeutic management of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years, remaining at the intensive care of the Saint-Luc University Hospital
* Recently transferred from emergency care with Community acquired Pneumonia of grade 4 suspicion
* With a Ventilation acquired Pneumonia suspicion

Suspicion will be based on symptoms, clinical, biological and radiological criteria.

Exclusion Criteria:

* Patients from whom no respiratory sample can be obtained
* Patients benefitting from palliative care
* Insufficient volume of the respiratory sample after routine testing to perform the FA-PNEU test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Turn Around Time Treatment | 48 hours from arrival of the respiratory sample at the laboratory
  Turn Around Time administration of optimal antimicrobial treatment

SECONDARY OUTCOMES:
Performances FilmArray Pneumonia | 1 week from arrival of the respiratory sample at the laboratory
  Microbiological performances FA-PNEU test versus routine microbiology testing

CONTACTS AND LOCATIONS:
Overall Officials: Alexia VERROKEN, Principal Investigator — Cliniques universitaires St-Luc
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerneis S, Visseaux B, Armand-Lefevre L, Timsit JF. Molecular diagnostic methods for pneumonia: how can they be applied in practice? Curr Opin Infect Dis. 2021 Apr 1;34(2):118-125. doi: 10.1097/QCO.0000000000000713. PMID 33395094